CLINICAL TRIAL: NCT00327535
Title: A Multicenter, Randomized, Open Label Dose Finding Study of Mircera in Anemic Patients With Stage IIIB or IV Non-small Cell Lung Cancer Receiving First Line Myelosuppressive Chemotherapy
Brief Title: A Study of Mircera in Anemic Patients With Non-Small Cell Lung Cancer Receiving First Line Chemotherapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH19960
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa; continuous erythropoietin receptor activator

ARMS (4):
- Mircera 6.3 micrograms/kg (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Mircera 9 micrograms/kg (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Mircera 12 micrograms/kg (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — According to the approved local label (6.75 micrograms/kg every 3 weeks, or 2.25 micrograms/kg every week)
  Arms: Darbepoetin alfa
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 6.3 micrograms/kg every 3 weeks
  Arms: Mircera 6.3 micrograms/kg
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 9 micrograms/kg every 3 weeks
  Arms: Mircera 9 micrograms/kg
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 12 micrograms/kg every 3 weeks
  Arms: Mircera 12 micrograms/kg

SUMMARY:
This 4 arm study will assess the optimal starting dose of Mircera in the treatment of anemia in patients with non-small cell lung cancer receiving first line myelosuppressive chemotherapy. Patients will be randomized to receive either Mircera 6.3 micrograms/kg, 9 micrograms/kg or 12 micrograms/kg s.c. every 3 weeks or darbepoetin alfa according to the approved local label (either 6.75 micrograms/kg s.c. every 3 weeks, or 2.25 micrograms/kg every week). The anticipated time on study treatment is <3 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age;
* stage III or IV non-small cell lung cancer receiving first line myelosuppressive chemotherapy;
* myelosuppressive chemotherapy scheduled for at least 9 weeks;
* anemia at screening visit.

Exclusion Criteria:

* transfusion of red blood cells during the 4 weeks prior to first planned dose of study medication;
* iron deficiency anemia, or anemia caused by gastrointestinal bleeding;
* prior treatment with Mircera.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Average Hb change from baseline | Weeks 5-13

SECONDARY OUTCOMES:
Target Hb therapeutic range, average Hb values, hematopoietic response. | Days 2-85
Red blood cell (RBC) transfusions | Weeks 5-13
Adverse events (AEs), laboratory parameters, premature withdrawals | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (59):
- Australia (3):
  - East Bentleigh
  - Kurralta Park
  - Milton
- Austria (3):
  - Linz
  - Salzburg
  - Vienna
- Belgium (3):
  - Aalst
  - Edegem
  - Liège
- Toronto, Ontario, Canada
- Czechia (4):
  - Brno
  - Hradec Králové
  - Ostrava
  - Prague
- Estonia (2):
  - Tallinn
  - Tartu
- Helsinki, Finland
- France (8):
  - Bobigny
  - Caen
  - Dijon
  - Lyon
  - Paris
  - Pessac
  - Pierre-Bénite
  - Saint-Pierre
- Germany (5):
  - Gauting
  - Hamburg
  - Heidelberg
  - Karlsruhe
  - Trier
- Greece (4):
  - Athens
  - Heraklion
  - Larissa
  - Thessaloniki
- Hong Kong, Hong Kong
- Hungary (5):
  - Budapest
  - Deszk
  - Mátraháza
  - Nyíregyháza
  - Székesfehérvár
- Italy (7):
  - Genova
  - Legnago
  - Novara
  - Pavia
  - Ravenna
  - San Giovanni Rotondo
  - Sassari
- Poland (7):
  - Bydgoszcz
  - Elblag
  - Otwock
  - Poznan
  - Radom
  - Wroclaw
  - Włocławek
- Spain (5):
  - Barcelona
  - Girona
  - Madrid
  - San Cristóbal de La Laguna
  - Zaragoza